CLINICAL TRIAL: NCT06410443
Title: Efficacy and Safety of Local Glucocorticoids for the Treatment of Acute Radiation-Induced Intestinal Injury: A Randomized Controlled Trial
Brief Title: Efficacy and Safety of Local Glucocorticoids for the Treatment of Acute Radiation-Induced Intestinal Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Xingshun Qi, Director of Department of Gastroenterology, General Hospital of Shenyang Military Region
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XHNKKY-RII-RCT
Record Dates: First submitted 2024-04-30; First posted 2024-05-13 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Radiation-Induced Intestinal Injury
Keywords: Radiation-Induced Intestinal Injury; glucocorticoid
MeSH Terms: interventions — Dexamethasone; Anti-Bacterial Agents; Probiotics; Vitamins; Antidiarrheals; Enteral Nutrition

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glucocorticoids+routine treatment group (Experimental): Dexamethasone retention enema
  Interventions: Drug: Dexamethasone; Drug: Antibiotics, probiotics, vitamins, antidiarrheal drugs, enteral nutrition, and endoscopic argon plasma coagulation
- Routine treatment group (Active Comparator): Routine treatment of acute radiation-induced intestinal injury according to the current practice guideline
  Interventions: Drug: Antibiotics, probiotics, vitamins, antidiarrheal drugs, enteral nutrition, and endoscopic argon plasma coagulation

INTERVENTIONS:
Drug: Dexamethasone — Retention enema with 10mg dexamethasone, once a day, the total course of treatment for 1 week.
  Other Names: RHP
  Arms: Glucocorticoids+routine treatment group
Drug: Antibiotics, probiotics, vitamins, antidiarrheal drugs, enteral nutrition, and endoscopic argon plasma coagulation — Treatment according to guideline of radiation-induced intestinal injury.

SUMMARY:
Due to the increasing number and prolonged survival of malignant tumor patients treated with radiotherapy, the complication, such as acute radiation-induced intestinal injury, has become increasingly significant. Glucocorticoids may play a therapeutic role by regulating the inflammatory response in patients with acute radiation-induced intestinal injury. However, the conclusions of related studies were controversial.

DETAILED DESCRIPTION:
A total of 60 patients with acute radiation-induced intestinal injury will be enrolled. They will be randomly assigned at a 1:1 ratio into glucocorticoid group and standard treatment group. The primary endpoint is the recovery and improvement of acute radiation-induced intestinal injury. The secondary study endpoints include the recurrence and aggravation of radiation-induced intestinal injury, and adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Grade II-III acute radiation-induced rectosigmoid injury
2. Signed informed consents
3. Age ≥18 years
4. Rstimated survival time >1 year

Exclusion Criteria:

1. Absolute contraindications to glucocorticoids
2. A history of glucocorticoids treatment within 3 months
3. Inflammatory bowel disease or infectious intestinal disease
4. Recurrence of malignant tumor
5. Colorectal cancer or metastasis
6. Severe heart or lung diseases
7. Recent history of surgery or trauma
8. Poorly controlled hyperglycemia and hypertension
9. Active tuberculosis
10. Ssevere gastrointestinal ulcers
11. Glaucoma
12. Sychiatric diseases
13. Pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Recovery and/or improvement | 3 months
  1. If patients' clinical symptoms, including abdominal pain, diarrhea, and hematochezia, and intestinal mucosal lesions under endoscopy disappear, the recovery will be defined.
  2. If patients' clinical symptoms alleviate, and/or the Vienna scores evaluated by endoscopy decrease at least 1 point, the improvement will be defined.
  The total number and frequency of patients who have both recovery and improvement of radiation-induced intestinal injury after treatment is calculated as the treatment efficacy.

SECONDARY OUTCOMES:
Recurrence and/or aggravation | 1 year
  Clinical symptoms related to radiation-induced intestinal injury and intestinal mucosal lesions under endoscopy recur or aggravate.
Adverse events | 1 year
  Any adverse event develop.

CONTACTS AND LOCATIONS:
Overall Officials: Xingshun Qi, Principal Investigator — The General Hospital of Northern Theater Command; Xiaofeng Liu, Principal Investigator — The 960th Hospital of the Chinese People's Liberation Army; Xiaohua Bao, Principal Investigator — The 964th Hospital of the Chinese People's Liberation Army; Cheng Bai, Principal Investigator — The 967th Hospital of the Chinese People's Liberation Army; Junchen Ge, Principal Investigator — The 962rd Hospital of the Chinese People's Liberation Army; Dongshuai Su, Principal Investigator — The 963rd Hospital of the Chinese People's Liberation Army; Wenda Xu, Principal Investigator — The 81th Group Military Hospital of of the Chinese People's Liberation Army; Ran Jiang, Principal Investigator — The 966th Hospital of the Chinese People's Liberation Army; Yumei Hou, Principal Investigator — 92493 Hospital of the Chinese People's Liberation Army; Hong Dai, Principal Investigator — Liaoning Provincial Corps Hospital of the Chinese People's Armed Police; Bingguo Piao, Principal Investigator — The 78th Group Military Hospital of the Chinese People's Liberation Army; Yufeng Zhang, Principal Investigator — The 79th Group Military Hospital of of the Chinese People's Liberation Army; Lichun Shao, Principal Investigator — Air Force Hospital of Northern Theater Command; Haijun Liang, Principal Investigator — 96605 Hospital of the Chinese People's Liberation Army
Locations (1):
- Department of Gastroenterology, General Hospital of Northern Theater Command (formerly called General Hospital of Shenyang Military Area), Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kochhar R, Patel F, Dhar A, Sharma SC, Ayyagari S, Aggarwal R, Goenka MK, Gupta BD, Mehta SK. Radiation-induced proctosigmoiditis. Prospective, randomized, double-blind controlled trial of oral sulfasalazine plus rectal steroids versus rectal sucralfate. Dig Dis Sci. 1991 Jan;36(1):103-7. doi: 10.1007/BF01300096. PMID 1670631
- [Result] Chen W, Ma Q, Yang L, Zhang L, Zhu J, Lin W. Curative effects of montmorillonite powder combined with dexamethasone on acute radiation enteritis. Am J Transl Res. 2021 Jun 15;13(6):7270-7275. eCollection 2021. PMID 34306492
- [Derived] Li Q, Liu X, Shao L, Bao X, Bai C, Ge J, Su D, Xu W, Jiang R, Mu Z, Dai H, Piao B, Zhang Y, Liang H, Yan Y, Zhang C, Xu X, Chen J, Wang J, Zhang J, Zhang J, Zhang Y, Wang J, Yang Q, Li X, Zhang X, Hou Y, Jiang R, Jin H, Qi X, Wang H. Efficacy and safety of local glucocorticoids for the treatment of acute radiation-induced intestinal injury: protocol of a multicenter randomized controlled trial. Front Pharmacol. 2025 May 30;16:1529977. doi: 10.3389/fphar.2025.1529977. eCollection 2025. PMID 40520206